CLINICAL TRIAL: NCT07289074
Title: Neurokinin A and Matrix Metalloproteinase 9 Levels in Gingival Crevicular Fluid Samples of Teeth With Symptomatic Irreversible Pulpitis With Symptomatic Apical Periodontitis: A Comparative Cross Sectional Study
Brief Title: Neurokinin A and Matrix Metalloproteinase 9 Levels in Gingival Crevicular Fluid Samples of Teeth With Symptomatic Irreversible Pulpitis With Symptomatic Apical Periodontitis
Status: Not yet recruiting | Type: Observational
Sponsor: Hadeer Mostafa El Mohamady El Feky (Other)
Responsible Party: Sponsor-Investigator, Hadeer Mostafa El Mohamady El Feky, PhD Candidate at Faculty of Dentistry- Endodontic Department (Cairo univerity), Cairo University
Organization: Cairo University (Other)
Other Study IDs: Hadeer Mostafa -14422022580639
Record Dates: First submitted 2025-11-25; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Symptomatic Irreversible Pulpitis With Apical Peridontitis
Keywords: Gingival crevicular fluid; Matrix Metalloproteinase 9; Neurokinin A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with symptomatic irreversible pulpitis with symptomatic apical peridontitis: * Gingival crevicular fluid samples will be collected from the symptomatic teeth and from the healthy contalateral teeth with normal pulp to detect the lavel of Neurokinin A (NKA) and Matrix metalloproteinase-9 (MMP-9) in the diseased teeth and compare it with that of the healthy teeth.
  * The study will also correlate the level of these biomarkers with the preoperative pain severity using the Numerical Rating Scale (NRS).
  Interventions: Diagnostic Test: Gingival crevicular fluid samples from the symptomatic teeth and the healthy contrlateral teeth
- The healthy contralateral teeth of tha same patients: * Gingival crevicular fluid samples will be collected from the symptomatic teeth and from the healthy contalateral teeth to detect the lavel of Neurokinin A (NKA) and Matrix metalloproteinase-9 (MMP-9) in the diseased teeth and compare it with that of the healthy contralateral teeth.
  * The study will also correlate the level of these biomarkers and the preoperative pain severity using the Numerical Rating Scale (NRS).
  Interventions: Diagnostic Test: Gingival crevicular fluid samples from the symptomatic teeth and the healthy contrlateral teeth

INTERVENTIONS:
Diagnostic Test: Gingival crevicular fluid samples from the symptomatic teeth and the healthy contrlateral teeth — The detection of the inflammatory biomarkers levels in the gingival crevicular fluid of the symptomatic teeth is considered an objective,molecular-based and non invasive method for diagnosis.
  Other Names: Matrix Metalloproteinase 9 and Neurokinin A will be detected in gingival crevicular fluid samples by using ELISA kits; correlate the level of these diagnostic biomarkers with the pre-operative pain severity by using the numerical rating scale

SUMMARY:
The aim of this study is to investigate the levels Neurokinin A and of Matrix Mtalloproteinase (MMP-9) in gingival crevicular fluid samples (GCF) as potential biomarkers for the diagnosis of symptomatic irreversible pulpitis with symptomatic apical periodontitis and to correlate the level of these diagnostic biomarkers ( Nerokinin A and MMP-9) with the pre-operative pain severity using the Numerical Rating Scale (NRS).

This study will utilize a comparative cross-sectional design to assess the levels of Neurokinin A (NKA) and Matrix metalloproteinase-9 (MMP-9) in gingival crevicular fluid (GCF) samples from symptomatic and healthy contralateral teeth with normal pulp.

DETAILED DESCRIPTION:
The study design is Comparative Cross sectional study. The study will be conducted at the Dental hospital of Cairo University with access to patients undergoing treatment for teeth with pulpitis and apical periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18-60) diagnosed with symptomatic irreversible pulpitis with symptomatic apical periodontitis and have healthy contralateral teeth with normal pulp.
* The involved teeth should have healthy periodontal conditions (Normal periodontal pocket depth, No bleeding on Probing and No mobility).
* Patients who have not undergone any previous dental treatments in the involved teeth.
* Signed informed consent.

Exclusion Criteria:

* Patients with systemic diseases affecting the immune response (e.g., autoimmune diseases, uncontrolled diabetes).
* Patients taking medications that can affect the inflammatory markers (e.g., Steroids and Tetracyclins).
* Smokers.
* Individuals with periodontal disease unrelated to apical periodontitis.
* Presence of marginal bone loss.
* Pregnant women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults (aged 18-60) diagnosed with symptomatic irreversible pulpitis with symptomatic apical periodontitis and have their healthy contralateral teeth with normal pulp with clinically healthy periodontium and not undergone any previous treatments in the involved teeth.
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The level of Neurokinin A in gingival crevicular fluid samples of teeth diagnosed with symptomatic irreversible pulpitis with symptomatic apical peridontitis and the contralateral teeth with healthy normal pulp. | Pre-operative measurement for Neurokinin A in gingival crevicular fluid samples
  Method of Measurement:
  Human Neurokinin A ELISA Kit (Bioassay Technology Laboratory, Shanghai, China) - Unit of measurement: Pg/ml

SECONDARY OUTCOMES:
A- The level of MMP-9 in gingival crevicular fluid samples of the symptomatic teeth and the contralateral teeth with normal pulp. B- The pre-operative pain severity in relation with the levels of these diagnostic biomarkers (Nerokinin A and MMP-9). | A- Pre-operative measurement for Matrix Metalloproteinase 9 in gingival crevicular fluid samples. B- Pre-operative pain severity assessment to corelate it with the levels of these diagnostic biomarkers (Nerokinin A and MMP-9)..
  Methods of measurement:
  A- Human Matrix Metalloproteinase 9;Gelatinase B- ELISA Kit: (Bioassay Technology Laboratory, Shanghai, China) - Unit of measurement: Pg/ml
  B- The Numerical Rating Scale (NRS): is a commonly used tool for assessing pain severity and consists of a line (either vertical or horizontal) divided into 11 numbers ranging from 0 to 10, where 0 represents no pain and 10 represents the worst possible pain - Unit of measurement: Score (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Saied M Abdel Aziz, Professor of Endodontics, Study Director — Faculy of Dentistry, Cairo university, Egypt
Locations (1):
- Faculty of Dentistry, Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No